CLINICAL TRIAL: NCT04082741
Title: A Phase 1, Double-Blind, Placebo-Controlled, Randomized Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Exploratory Pharmacodynamics of Oral BMS-986318 Administration in Healthy Participants
Brief Title: A Single and Multiple Ascending Dose Study of BMS-986318 in Healthy Participants
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: The study is no longer required based on nonclinical drug data
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IM031-002
Record Dates: First submitted 2019-08-15; First posted 2019-09-09 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Healthy Participants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monotherapy SAD BMS-986318 or Placebo (Experimental): Single Ascending Dose (SAD)
  Interventions: Drug: BMS-986318; Other: Placebo
- Monotherapy MAD BMS-986318 or Placebo (Experimental): Multiple Ascending Dose (MAD)
  Interventions: Drug: BMS-986318; Other: Placebo

INTERVENTIONS:
Drug: BMS-986318 — Specified dose on specified days
Other: Placebo — Placebo Matching BMS-986318

SUMMARY:
A study to evaluate single and multiple ascending doses of experimental medicine BMS-986318 in healthy participants.

DETAILED DESCRIPTION:
A Phase 1, Double-Blind, Placebo-Controlled, Randomized Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Exploratory Pharmacodynamics of Oral BMS-986318 Administration in Healthy Participants

ELIGIBILITY:
Inclusion Criteria:

* Healthy Participants as determined by no clinically significant deviations from normal in medical history, physical examination, ECG and clinical laboratory results as determined by the investigator
* Male participants who are sexually active with Women of Child Bearing Potential (WOCBP) must agree to follow instructions for methods of contraception for duration of treatment plus 92 days.
* Female participants must have documented proof that they are not of childbearing potential and a negative pregnancy test at screening and within 24 hours before the first dose of study treatment.

Exclusion Criteria:

* Use of any prescription drugs within 4 weeks or use of over-the-counter (OTC) medications or herbal preparations within 2 weeks prior to study treatment administration (except acid controllers, which are not allowed within 4 weeks prior to study treatment administration
* Women of Child Bearing Potential (WOCBP) or women who are breastfeeding.
* Any major surgery within 12 weeks of study administration Or any history of GI surgeries as listed.(eg, gastric bypass, gastric banding, Roux-en-Y) or gastric- emptying issues that could impact upon the absorption of nutrients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07-18 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Incidence of non-serious adverse events (AEs) | up to 30 days
Incidence of Serious Adverse Events (SAE) | up to 30 days
Incidence of AEs leading to discontinuation of study treatment | up to 30 days
Physical Examination of height | up to 30 days
Physical Examination of weight | up to 30 days
Physical Examination of BMI | up to 30 days
Assessment of body temperature | up to 30 days
Assessment of respiratory rate | up to 30 days
Assessment of blood pressure | up to 30 days
Number of participants with 12-lead Electrocardiogram (ECG) Abnormalities | up to 30 days
Number of clinical significant changes in lab assessment of blood serum | up to 30 days
Number of Clinically significant changes in assessment of blood | up to 30 days
Number of Clinically significant changes in lab assessment of urine | up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PRA Health Sciences - Lenexa, Lenexa, Kansas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/investigator-inquiry-form.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm